CLINICAL TRIAL: NCT04062097
Title: Registration of Idarucizumab for Patients with IntraCranial Hemorrhage (RIC-ICH)
Brief Title: Registration of Idarucizumab for Patients with IntraCranial Hemorrhage
Acronym: RIC-ICH
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hans Diener, Senior Professor of Clinical Neurosciences, University Hospital, Essen
Other Study IDs: RIC-ICH
Record Dates: First submitted 2019-08-08; First posted 2019-08-20 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2022-04

CONDITIONS: Intracranial Hemorrhage
Keywords: intracranial/intracerebral bleeding; stroke; transient ischemic attack (TIA); myocardial infarction; anticoagulation; dabigatran; idarucizumab; vitamin-k antagonists
MeSH Terms: conditions — Intracranial Hemorrhages; Stroke; Ischemic Attack, Transient; Myocardial Infarction | interventions — Dabigatran; idarucizumab; acarboxyprothrombin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- dabigatran-group: Patients with the anticoagulating therapy dabigatran and onset of clinically symptomatic intracranial hemorrhage, that is treated with idarucizumab.
  Interventions: Drug: Dabigatran Etexilate Oral Capsule [Pradaxa]; Drug: Idarucizumab 2.5 GM/50 ML Intravenous Solution [PRAXBIND]
- VKA-group: Patients under effective treatment with VKA and with intracranial hemorrhage.
  Interventions: Drug: Vitamin K antagonist

INTERVENTIONS:
Drug: Dabigatran Etexilate Oral Capsule [Pradaxa] — Dabigatran is the most frequently used direct thrombin inhibitor in secondary stroke prevention in patients with atrial fibrillation.
  Groups: dabigatran-group
Drug: Idarucizumab 2.5 GM/50 ML Intravenous Solution [PRAXBIND] — Idarucizumab is the current standard therapy in patients with intracranial bleeding under anticoagulation with dabigatran.
  Groups: dabigatran-group
Drug: Vitamin K antagonist — This drug group includes the active substances phenprocoumon and warfarin.
  Groups: VKA-group

SUMMARY:
This multicenter, prospective, observational, non-interventional study investigates patients with intracranial hemorrhage under effective anticoagulation with dabigatran or vitamin-K antagonist (VKA). Routine data will be collected during hospitalization. Patients aged 18 years or older under effective therapy with dabigatran and symptomatic intracranial bleeding confirmed by cerebral imaging and treated with idarucizumab will be compared to patients under effective treatment with VKA at the time of onset of the intracranial bleeding. Ninety-five dabigatran patients who provided written informed consent for data transmission will be included. As control group retrospective and anonymized data of 285 VKA patients patients under VKA treatment and admitted to RIC-ICH study centers will be used. For each patient receiving idarucizumab, three patients with intracranial hemorrhage under effective treatment with VKA, will be included (retrospective) in the study. In addition, data of VKA patients will be transferred from the RASUNOA-PRIME and the "Erlanger Hirnblutungs-Register".

ELIGIBILITY:
Inclusion Criteria (dabigatran-group):

* Age ≥18 years at enrollment
* Patients willing and able to provide written informed consent for data transmission (exceptions/special cases for patients who are not legally competent to sign informed consent for data transmission).
* Patients with primary intracranial hemorrhage as confirmed with CT.
* Patients under effective anticoagulation treatment with dabigatran at the time of admission (TT>60 sec. or last intake of medication <24hours).
* Patients treated with Idarucizumab (2x2.5 g recommended) may still be included the day after the administration of Praxbind, or on the following working day if treatment was carried out on the weekend.
* inclusion (signed informed consent) as soon as possible after start of symptoms of initial ICH event, but before discharge.

Inclusion Criteria (control-group):

- Patients with intracranial hemorrhage under effective anticoagulation treatment with VKA (INR ≥ 1,7) having been initially treated in the past in the study center.

Exclusion Criteria (dabigatran-group):

* Additional therapy with PCC, aPCC or factor VII (in patients under dabigatran).

Exclusion Criteria (all patients):

- Start of symptoms of initial ICH event > 24 h before admission to hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the anticoagulating therapy dabigatran admitted with a clinically symptomatic intracranial bleeding will be included in the study, if they have been treated with idarucizumab (dabigatran-group). It is assumed that some of these patients will have been given an antiplatelet drug as co-medication.
  As reference population, patients with intracranial hemorrhage under effective treatment with VKA (INR ≥ 1,7) treated in the same center will be used (VKA-group). These patients usually have been treated with some antagonist to VKA (or no reversal therapy at all).
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Intra-hospital mortality rate | From study inclusion until hospital discharge or 30 days after index event, whichever came first.
  Intra-hospital mortality rate

SECONDARY OUTCOMES:
Change in National Institutes of Health Stroke Scale (NIHSS) | At hospital admission, 24 hours after admission and 72 hours after admission.
  Change in National Institutes of Health Stroke Scale (NIHSS) of ≥4 pts compared to initial NIHSS or worsening of NIHSS level of consciousness ≥1 point or increase of the volume of the intracranial bleeding or new intraventricular bleeding or death. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Intracranial bleeding | Between 24 and 72 hours after initial CT.
  Change in size/volume of > 33% or ≥ 6.5 ml of the intracranial bleeding evaluated by first CT
Stroke severity | 72 hours after hospital admission
  Change in stroke severity by ≥4 points based on National Institutes of Health Stroke Scale (NIHSS). The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Functional status | At hospital discharge or 30 days after index event, whichever came first.
  Functional status according to modified Rankin Scale (mRS). The scale runs from 0-6, running from perfect health without symptoms to death: 0 - No symptoms, 1 - No significant disability, 2 - Slight disability, 3 - Moderate disability, 4 - Moderately severe disability, 5 - Severe disability, 6 - Dead.
Mortality rate | 7 and 30 days after index event.
  Mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Hans Diener, Prof. Dr., Study Director — University Hospital, Essen
Locations (33):
- Germany (33):
  - Klinikum Schön Klinik Bad Aibling SE & Co. KG, Bad Aibling
  - Hochtaunuskliniken GmbH, Bad Homburg
  - Rhön Klinikum Campus Bad Neustadt, Bad Neustadt an der Saale
  - Vivantes Klinikum Auguste Viktoria, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Vivantes Humboldt Klinikum, Berlin
  - Evangelisches Klinikum Bethel gGmbH, Bielefeld
  - Katholisches Klinikum Bochum gGmbH, St. Josef Hospital, Bochum
  - Universitätsklinkum Bonn, Bonn
  - Klinikum Allgemeines Krankenhaus Celle, Celle
  - Carl-Thiem-Klinikum Cottbus gGmbH, Cottbus
  - Krankenhaus St. Elisabeth gGmbH, Damme
  - Albert-Ludwigs-Universität Freiburg, Freiburg im Breisgau
  - SHR Wald-Klinikum Gera GmbH, Gera
  - Georg-August-Universität Göttingen, Universitätsmedizin, Göttingen
  - Klinikum Martha Maria, Halle
  - Asklepios Klinik Wandsbek, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum Agatharied GmbH, Hausham
  - Universitätsklinikum Heidelberg, Heidelberg
  - BDH-Klinik Hessisch Oldendorf, Hessisch Oldendorf
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universität Leipzig, Leipzig
  - Klinikum Main-Spessart Lohr, Lohr
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsmedizin der Johannes-Guttenberg-Universität Mainz, Mainz
  - Klinikum Osnabrück, Osnabrück
  - Klinikum Vest Knappschaftskrankenhaus, Recklinghausen
  - Klinikum Nordwest Krankenhaus Sande, Sanderbusch
  - Klinikum der Landeshauptstadt Stuttgart gKAöR, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
  - Sana HANSE-Klinikum Wismar GmbH, Wismar